CLINICAL TRIAL: NCT05617027
Title: Relieving Chronic Pain in Older Adults With Transcranial Direct Current Stimulation
Acronym: tDCS-pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-31-2022-4641
Record Dates: First submitted 2022-10-25; First posted 2022-11-15 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-07

CONDITIONS: Pain, Chronic
Keywords: Chronic pain; transcranial direct current stimulation; quality of life
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial (RCT) with placebo that includes two parallel groups (real tDCS and placebo tDCS), with random assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and team members, also referred to as evaluator members above (researchers, analysts, physical therapists, and research assistants) will all be blinded to the intervention, except for those not involved in data collection and analysis: a) the statistician who will generate the randomization list, b) the computer team who will program the randomization system, and c) the interventionist who will apply the tDCS power.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- actual tDCS (Experimental): The actual transcranial direct current stimulation (tDCS) intervention will be conducted by a physiotherapist who will perform 5 sessions of actual tDCS , 5 consecutive days, for 20 minutes of treatment for a total of 45 minutes at the clinic for each session.
  The tDCS current will be 2 mA for the whole 20-minute session.
  Interventions: Other: actual transcranial direct current stimulation (tDCS)
- placebo tDCS (Placebo Comparator): The placebo transcranial direct current stimulation (tDCS) intervention will be conducted by a physiotherapist who will perform 5 sessions of placebo tDCS, 5 consecutive days, for 20 minutes of treatment for a total of 45 minutes at the clinic for each session.
  The tDCS current will be 2 mA for 30 secondes, and then will strop for the rest of the 20-minute session (programming of the equipment).
  Interventions: Other: placebo transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Other: actual transcranial direct current stimulation (tDCS) — tDCS is a non-invasive brain stimulation technique that would influence the brain's pain control mechanisms.
  The anode is attached to the skull above the M1 opposite the painful side (in case of unilateral pain) or opposite the dominant hand (in case of bilateral pain). The cathode (at the supraorbital level opposite the stimulated M1) will be positioned using the 10-20 EEG system and the tDCS intensity will be 2 mA.
  Arms: actual tDCS
Other: placebo transcranial direct current stimulation (tDCS) — The anode is attached to the skull above the M1 opposite the painful side (in case of unilateral pain) or opposite the dominant hand (in case of bilateral pain). The cathode (at the supraorbital level opposite the stimulated M1) will be positioned using the 10-20 EEG system and the tDCS intensity will be 2 mA for 30 secondes, and then 0 mA for the rest of the 20-minute session.
  Arms: placebo tDCS

SUMMARY:
The primary objective of this study is to determine, in a healthcare setting, the effectiveness of actual tDCS in reducing pain compared with placebo tDCS. This is a multicenter randomized controlled trial with parallel groups (real tDCS vs. placebo) blinded to participants, assessors and tDCS providers. The real tDCS group will receive a daily 20-minute session of tDCS (current intensity = 2 mA), for 5 consecutive days, while the placebo tDCS group will receive an equivalent treatment, but the current will be stopped after the first 30 seconds. The study will take place in 5 rehabilitation clinics in 3 Quebec regions. One hundred and fifty (150) seniors aged 65 years or older with chronic (> 6 months), moderate to severe musculoskeletal pain will be recruited (50 participants/region). Follow-ups will take place at 1 week and 3 months post-treatment. The primary dependent variable is pain intensity (numerical scale from 0 to 10). Secondary variables will be measured using standardized and validated questionnaires: 1) pain-related interferences (physical function, mood, quality of life) and 2) perception of post-TDCS changes. Neurophysiological measures (pain control pathways).

DETAILED DESCRIPTION:
Rationale : Chronic pain is the leading cause of disability and affects a large number of seniors. Transcranial direct current stimulation (tDCS), which provides non-invasive stimulation of the brain, is a promising avenue for relieving pain that is refractory to traditional treatments. To date, however, its clinical efficacy has yet to be confirmed in the elderly.

Objectives : The primary objective of this study is to determine, in a healthcare setting, the effectiveness of actual tDCS in reducing pain compared with placebo tDCS. Secondary objectives are to assess the effect of tDCS on pain-related interference and the relationship between the response to tDCS and the integrity of pain control systems (descending pathways controlling pain circuits).

Methods : This is a multicenter randomized controlled trial with parallel groups (real tDCS vs. placebo) blinded to participants, assessors and tDCS providers. The real tDCS group will receive a daily 20-minute session of tDCS (current intensity = 2 mA), for 5 consecutive days, while the placebo tDCS group will receive an equivalent treatment, but the current will be stopped after the first 30 seconds. The study will take place in 5 rehabilitation clinics in 3 Quebec regions: Sherbrooke (n=1), Quebec City (n=2), Montreal (n=2). One hundred and fifty (150) seniors aged 65 years or older with chronic (> 6 months), moderate to severe musculoskeletal pain will be recruited (50 participants/region). Follow-ups will take place at 1 week and 3 months post-treatment. The primary dependent variable is pain intensity (numerical scale from 0 to 10). Secondary variables will be measured using standardized and validated questionnaires: 1) pain-related interferences (physical function, mood, quality of life) and 2) perception of post-TDCS changes. Neurophysiological measures (pain control pathways), i.e., the integrity of corticothalamic and corticospinal projections will be tested by diffusion MRI and transcranial magnetic stimulation.

Anticipated results: Our hypotheses are that (i) real tDCS will be more effective in reducing pain intensity than placebo tDCS at 1 week post-treatment. This reduction in pain will be maintained at the 3-month post-treatment follow-up of real tDCS. (ii) Real tDCS will be more effective than placebo treatment in reducing pain interference with physical function, mood and quality of life. Perceived improvement with the treatment received will also be greater for real tDCS. (iii) Individuals with stronger cortico-thalamic and corticospinal projections in pre-tDCS will be more relieved by actual tDCS than those with less strong projections.

Ultimately, this study will allow us to evaluate the effectiveness of tDCS in the care setting for the relief of chronic musculoskeletal pain in the elderly and to identify those individuals most likely to respond to this type of treatment based on potential biomarkers related to the integrity of the pain control system.

ELIGIBILITY:
Inclusion Criteria:

* Be aged ≥ 65 years
* Have chronic (≥ 6 months) musculoskeletal pain of moderate to severe intensity (≥4 out of 10 on a numerical scale of 0 to 10)

Exclusion Criteria:

* Those with contraindications to tDCS
* Those with contraindications to TMS
* Those with contraindications to IRM
* Individuals for whom the procedure could cause impairment of well-being, or has another medical condition that could put them at risk in the judgment of a health care professional.
* Patients taking medications that act on the GABAergic and glutamatergic systems (modulating tDCS effects) will be excluded
* Individuals taking other types of medications or receiving rehabilitation are not excluded but will be asked, in the absence of clinical contraindication, to avoid any modification (e.g., new treatment, discontinuation, or change in dose) during the study.
* People with epilepsy and seizures will not be excluded from the study. The research team will simply be asked to pay closer attention to these participants during the administration of MST.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity from baseline to 1 week after the intervention | Mean of Patient reported pain on 5 consecutive days: i. 1 week before the intervention compared to1 week after the intervention
  Visual analogue scale (0-10) where 0 = no pain, 10= worst pain
Maintenance of the effect on pain after from to 1 week to 3 months after intervention | Mean of Patient reported pain on 5 consecutive days: 3 months after the intervention to see if the effect of the treatment is maintained.
  Visual analogue scale (0-10) where 0 = no pain, 10= worst pain

SECONDARY OUTCOMES:
Sociodemographic, life habits, and medical history data | Selection visit (pre-intervention)
  Questionnaire including questions regarding age, sex, gender, education, salary, drug use, coffee, tobacco, alcohol, diagnosis, time since onset of symptoms, concomitant medication.
Change in affective component of pain from baseline to 1 week and 3 months after intervention | i. 1 week before the intervention, ii. 1 week after the intervention, and iii. 3 months after the intervention
  McGill-Melzack Questionnaire: The 20 questions in this tool focus on the qualitative aspect of pain, for a total of 78 points, and are divided into 4 subcategories: sensory, affective, evaluative and miscellaneous. Higher is the score, the greater is the pain.
Change in mood from baseline to 1 week and 3 months after intervention | i. 1 week before the intervention, ii. 1 week after the intervention, and iii. 3 months after the intervention
  Hospital Anxiety and Depression Scale (HADS): 14-item questionnaire measured with a 4-point Likert scale (0 = no to 3 = yes, definitively). Higher score indicating higher distress.
Change in physical function related to pain from baseline to 1 week and 3 months after intervention | i. 1 week before the intervention, ii. 1 week after the intervention, and iii. 3 months after the intervention
  Brief Pain Inventory - short form (BPI): this 9 item questionnaire is use to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. It uses a 0 to 10 numeric rating scales for item rating. The BPI has no scoring algorithm.
Change in quality of life covering eight domains of health from baseline to 1 week and 3 months after intervention | i. 1 week before the intervention, ii. 1 week after the intervention, and iii. 3 months after the intervention
  36-Item Short Form Survey (SF-36): This questionnaire covers eight domains of health related to quality of life: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. A high score defines a more favorable health state.
Change in perception of change with treatment from 1 week to 3 months after intervention | i. 1 week after the intervention, and ii. 3 months after the intervention
  Patient Global Impression of Change (PGIC). This questionnaire assesses perceived changes using a 7-point scale, ranging from "Significantly Worsened" to "Significantly Improved.
Neurophysiological measures (MRI, Tractography) | i. 1 week before the intervention
  Magnetic resonance imaging (MRI) is an imaging test that uses powerful magnetic forces, radio waves and a computer to produce detailed 3-dimensional images of organs, bones and soft tissue inside your body. In this particular context, IRM will allow to quantify the integrity and morphology of myelinated corticospinal projection (in the brain) via a diffusion MRI and mathematical reconstruction of the tract (tractography analysis).
Functional neuroanatomical measurement (TMS) | i. 1 week before the intervention
  Transcranial Magnetic Stimulation (TMS): allows the evaluation of corticospinal projections. This technique aims to stimulate certain nerve cells via short magnetic pulses directed to the brain.This stimulation release a potential.known as a motor evoked potential, MEP which is then recorded using electromyography (EMG). The magnitude of muscle activity generated for a given TMS pulse strength forms a measure of cortical excitability in the stimulated region.

CONTACTS AND LOCATIONS:
Overall Officials: Guillume Léonard, Principal Investigator — Université de Sherbrooke
Locations (3):
- Canada (3):
  - Institut universitaire sur la réadaptation en déficience physique de Montréal (IURDPM), Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - Centre de recherche sur le vieillissement (CdRV), Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided